CLINICAL TRIAL: NCT02390570
Title: Incorporating Patient Capacity Into the Clinical Landscape
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kasey R. Boehmer, Health Services Analyst, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 14-008621
Record Dates: First submitted 2015-02-19; First posted 2015-03-17 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Chronic Disease
Keywords: Patient Capacity
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Implementation Arm (Experimental)
  Interventions: Other: Patient Capacity Assessment Instrument

INTERVENTIONS:
Other: Patient Capacity Assessment Instrument — The Patient Capacity Assessment instrument is a conversational tool designed to help patients and clinicians discuss capacity in clinicial conversations of primary care.

SUMMARY:
This study is designed to answer why "patient capacity" (i.e. patient available abilities and resources to enact self-care and access healthcare) is not regularly documented in the Electronic Medical Record (EMR) in a way that is useful for clinicians.

Through the implementation of communication tools designed for patient capacity assessment and engagement of stakeholders in a process of user-centered design, the study team hypothesizes that the study can help clinicians elicit this information in conversation and regularly document it in the medical record for future healthcare discussions.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have one or more chronic condition and do not have any barriers to consent (such as major cognitive disabilities) will be eligible for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-02-22 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Number of resource limitations measured by medical record review | Baseline up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Kasey Boehmer, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Boehmer KR, Dobler CC, Thota A, Branda M, Giblon R, Behnken E, Organick P, Allen SV, Shaw K, Montori VM. Changing conversations in primary care for patients living with chronic conditions: pilot and feasibility study of the ICAN Discussion Aid. BMJ Open. 2019 Sep 3;9(9):e029105. doi: 10.1136/bmjopen-2019-029105. PMID 31481553